CLINICAL TRIAL: NCT04871022
Title: Double-layer Versus Purse Uterine Closure Techniques : Impact on Residual Myometrial Thickness After Cesarean
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Ahmed Halouani, MD, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UTuniselmanar3
Record Dates: First submitted 2021-04-28; First posted 2021-05-04 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Uterine Scar Defect
Keywords: niche

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double layer unlocked uterine closer (Active Comparator): Double layer closure with a first continuous unlocked suture of the deep portion of the myometrium and a second unlocked continuous suture that approximate the upper portion of the myometrium.
  Interventions: Procedure: Double layer closure of the hysterotomy
- Purse uterine closer (Experimental): Purse suture of the uterus with a first continuous purse suture of the deep portion of the myometrium and a second unlocked continuous suture including the remaining part of the myometrium
  Interventions: Procedure: Purse closure of the hysterotomy

INTERVENTIONS:
Procedure: Double layer closure of the hysterotomy — Double layer closure with a first continuous unlocked suture of the deep portion of the myometrium and a second unlocked continuous suture that approximate the upper portion of the myometrium.
  Arms: Double layer unlocked uterine closer
Procedure: Purse closure of the hysterotomy — Purse suture of the uterus with a first continuous purse suture of the deep portion of the myometrium and a second unlocked continuous suture including the remaining part of the myometrium
  Arms: Purse uterine closer

SUMMARY:
There are different surgical techniques of uterine closure during cesarean. Currently data suggest that the double layer unlocked closure technique is associated with better uterine scar healing, and this technique is considered the gold standard.

This study compares two techniques of uterine closure on myometrium thickness:

1. Double layer unlocked suture;
2. Purse suture of the uterus with a first continuous purse suture of the deep portion of the myometrium and a second unlocked continuous suture including the remaining part of the myometrium.

The primary outcome is the mean residual myometrium thickness at the site of the uterine scar evaluated by transvaginal ultrasound at six months after cesarean.

ELIGIBILITY:
Inclusion Criteria:

* Planned cesarean
* Primary cesarean
* ≥ 38 gestational weeks

Exclusion Criteria:

* Previous cesarean
* Women < 18 years old
* Multiple gestation
* Mullerian anomalies
* Active labor
* Diabetes
* BMI >35 kg/m2
* Placenta praevia
* Chronic systemic disease
* Covid-19 infection

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Residual myometrium thickness | 6 months after intervention

SECONDARY OUTCOMES:
Operative time | Same day of intervention: day 1
Estimated blood loss | Same day of intervention: day 1
Mean number of haemostatic sutures | Same day of intervention: day 1
scar width | Same day of intervention: day 1

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital Mongi Slim la Marsa, Tunis, La Marsa, Tunisia

REFERENCES:
- [Derived] Halouani A, Dimassi K, Ben Mansour A, Triki A. Impact of purse-string uterine suture on scar healing after a cesarean delivery: a randomized controlled trial. Am J Obstet Gynecol MFM. 2023 Jul;5(7):100992. doi: 10.1016/j.ajogmf.2023.100992. Epub 2023 Apr 29. PMID 37127211